CLINICAL TRIAL: NCT03987087
Title: A Randomized Phase II Trial of Primary Tumor Radiotherapy for Patients With Malignant Pleural Effusion Stage IV Non-Small Cell Lung Cancer
Brief Title: A Randomized Study of Primary Tumor Radiotherapy for Patients With MPE Stage IV NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guizhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IV-NSCLC-MPE
Record Dates: First submitted 2019-06-12; First posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Malignant Pleural Effusion; Nonsmall Cell Lung Cancer, Stage IV
MeSH Terms: conditions — Pleural Effusion, Malignant; Carcinoma, Non-Small-Cell Lung | interventions — Radiation; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiotherapy group (Experimental): Thoracic intensity modulated radiation therapy (IMRT) concomitant with EGFR-TKI on paticipants with known sensitive EGFR mutations.Cisplatin Thoracenteral infusion chemotherapy。 Thoracic intensity modulated radiation therapy (IMRT) concomitant with Cisplatin Thoracenteral infusion chemotherapy and Systemic chemotherapy on paticipants with known NOT sensitive EGFR mutations.
  Interventions: Radiation: Radiation
- Chemotherapy group (Active Comparator): EGFR-TKI on paticipants with known sensitive EGFR mutations,Cisplatin Thoracenteral infusion chemotherapy.
  Cisplatin Thoracenteral infusion chemotherapy and Systemic chemotherapy on paticipants with known NOT sensitive EGFR mutations.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Radiation: Radiation — Thoracic intensity modulated radiation therapy (IMRT)
  +EGFR TKI combination Thoracenteral innfusion chemotherapy or Thoracenteral infusion chemotherapy combination Systemic chemotherapy
  Arms: Radiotherapy group
Drug: Chemotherapy — EGFR TKI combination Thoracenteral innfusion chemotherapy or Thoracenteral infusion chemotherapy combination Systemic chemotherapy
  Arms: Chemotherapy group

SUMMARY:
This randomized phase II study compare survival outcomes and toxicity of malignant pleural effusion stage IV non small-cell lung cancer patients Intrapleural infusion chemotherapy in combination with concurrent thoracic radiation therapy (TRT) VS not combination with concurrent thoracic radiation therapy (TRT).

DETAILED DESCRIPTION:
Malignant pleural effusion (MPE) is a common complication of stage IV NSCLC. MPE caused by lung cancer accounts for about 1/3. According to statistics, the number of MPE cases per year in the United States exceeds 150,000. At the same time, with the development of three-dimensional radiotherapy technology, the wide application of comprehensive treatment concept, and the understanding of the relationship between different metastatic state and survival of stage IV NSCLC, prospective and retrospective studies have confirmed that systemic therapy combined with primary tumor three-dimensional radiation Treatment is more conducive to improving symptoms and prolonging survival than medication alone. Retrospective results and prospective findings have been reported from the single center of the study group [Chinese Journal of Radiation Oncology, 2011, sixth issue and the first issue of 2012], taking local three-dimensional radical radiotherapy for chemotherapy, two Complementary technological advantages can significantly prolong survival and improve quality of life, enabling some patients to achieve long-term survival. However, most of the above studies excluded patients with malignant pleural effusion. For stage IV NSCLC of malignant pleural effusion, whether the primary tumor radiotherapy can bring survival benefits, has not yet formed a unified norm and conclusion, and needs further development. the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathological or cytological diagnosis, stage IV with malignant pleural effusion [UICC 2017 staging eighth edition] NSCLC patients;
* initial treatment (previously did not receive any treatment), it is recommended to complete the detection of driver genes (EGFR / ALK / ROS1) (tissue, blood);
* Age 18 to 80 years old, physical status score ECOG 0 to 2 or KPS ≥ 70 (see Annex 2); Metastatic lesions in the distant area: conscious when brain metastasis; the number of metastatic lesions in the lung does not affect lung function and may be treated with primary and/or partial metastases;
* no radiotherapy, EGFR-TKI and chemotherapy contraindications;
* primary tumor radiotherapy requires IMRT technology;
* Plan the design to give the primary tumor prescription dose (DTGTV) under the damage control threshold criteria;
* The planned dose includes 100% GTV, 90% of the prescribed dose includes 98%~100% of PTV [planned target dose (DTPTV)]; normal lung (full lung volume minus GTV volume) V20 ≤ 32%, MLD≤20Gy;
* metastatic tumor radiotherapy is a three-dimensional radiotherapy technique (IMRT/SRT/SBRT/VMAT, etc.), and large-segment radiotherapy.
* Subjects have no major organ dysfunction, or laboratory test indicators must meet the following requirements: Hematology: normal range according to laboratory standards; cardiac function: normal range; liver function: normal range; renal function: normal range Lung function: FEV1>50%, impaired light-moderate lung function.
* Informed consent (radiation, medication) before treatment;
* The patient has good compliance with the treatment and follow-up received.

Exclusion Criteria:

* Patients who do not meet the pathological type, stage, and survival status of the inclusion criteria;
* no malignant pleural effusion IV stage NSCLC;
* patients with malignant pericardial effusion; Diffuse liver metastasis, intrapulmonary metastasis and has seriously affected patients with liver and lung function;
* Patients with uncontrolled hypertension, diabetes, unstable angina, history of myocardial infarction, or symptomatic congestive heart failure or uncontrolled arrhythmias in the past 12 months; clinically diagnosed heart valve disease; • • •Active period of disease caused by bacteria, fungi or viruses; mental disorders; impaired severe lung function;
* pregnant, lactating patients;
* Patients with a history of other active malignancies other than small cell lung cancer before entering the group; non-melanoma skin basal cell carcinoma, in situ cervical cancer, and cured early prostate cancer;
* Patients with allergies and no known alternatives to known or suspected drugs in any study;
* Patients with poor compliance;
* Researchers believe that it is not appropriate to participate in this test.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival(PFS) | up to 9 months
  PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival(OS) | Time Frame: up to 9 months
  Overall survival is defined as the time interval from date of diagnosis to date of death from any cause Overall survival is defined as the time interval from date of diagnosis to date of death from any cause Overall survival is defined as the time interval from date of diagnosis to date of death from any cause Overall survival is defined as the time interval from date of diagnosis to date of death from any cause Overall survival is defined as the time interval from date of diagnosis to date of death from any cause
Treatment toxicities | Time Frame: up to 12 months
  To assess and record nausea, vomiting, hematologic toxicity,radiation oesophagitis and other treantment complications by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Guizhou Cancer Hospital, Guiyang, Guizhou, China

IPD SHARING:
Plan to Share IPD: Undecided